CLINICAL TRIAL: NCT03173300
Title: Clinical and Basic Investigations Into Phosphomannomutase Deficiency (PMM2-CDG)
Brief Title: Natural History Study Protocol in PMM2-CDG (CDG-Ia)
Status: Active, not recruiting | Type: Observational
Sponsor: Glycomine, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: GLY-000
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Phosphomannomutase 2 Deficiency
Keywords: PMM2-CDG; CDG-Ia
MeSH Terms: conditions — Congenital disorder of glycosylation type 1A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical and Basic Investigations into Phosphomannomutase deficiency (PMM2-CDG)

This is a natural history (observational) protocol designed to collect clinical and biological information in patients with PMM2-CDG (CDG-Ia).

DETAILED DESCRIPTION:
Subjects enrolled in this natural history study will be thoroughly examined for signs and symptoms of PMM2-CDG. Medical history, physical examination, laboratory testing and imaging studies will be performed during a single consultation. Follow-up will occur every 3- 6 months at a minimum, depending on the standard of care at the investigator's institution as well as the clinical status of the individual patient. All medical procedures are routine. No new therapy is offered as part of this study, and no change in the patients routine therapy is dictated by this protocol. The International Co-Operative Ataxia Rating Scale (ICARS) is to be performed every 3 months as an optional assessment. No randomization will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent/assent by the patient and/or their legally authorized representative
* Confirmed diagnosis of PMM2-CDG, based on enzymatic or molecular tests
* Willing and able to adhere to study requirements described in the protocol and consent/assent documents

Exclusion Criteria:

* Known or suspected differential diagnosis of any other known CDG (not PMM2-CDG)
* Currently using investigational drug
* Blood loss of ≥ 250 mL or donated blood within 56 days, or donated plasma within 7 days before study screening

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with PMM2-CDG, all ages
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-01-08 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Collect clinical and biological information in patients with CDG-PMM2 | up to 5 years
  Growth parameter, organ function tests, developmental tests, standard laboratory tests, disease severity score according to Nijmegen Paediatric CDG Rating Scale (NPCRS)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Glycomine, Inc.
Locations (11):
- United States (3):
  - Mayo Clinic College of Medicine, Rochester, Minnesota
  - Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington
- University Hospital Leuven, Leuven, Belgium, Belgium
- General University Hospital in Prague, Prague, Czechia
- Necker Enfants-Malades Hospital, Paris, France
- University Hospital of Catania, Catania, Italy
- Radboud University Nejmegen Medical Center, Nijmegen, Netherlands
- Mother and Child Institute (Instytut Matki i Dziecka), Warsaw, Poland
- Centro Hospitalar do Porto, Porto, Portugal
- Hospital Sant Joan de Déu, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pajusalu S, Vals MA, Serrano M, Witters P, Cechova A, Honzik T, Edmondson AC, Ficicioglu C, Barone R, De Lonlay P, Berat CM, Vuillaumier-Barrot S, Lam C, Patterson MC, Janssen MCH, Martins E, Quelhas D, Sykut-Cegielska J, Mousa J, Urreizti R, McWilliams P, Vernhes F, Plotkin H, Morava E, Ounap K. Genotype/Phenotype Relationship: Lessons From 137 Patients With PMM2-CDG. Hum Mutat. 2024 Oct 3;2024:8813121. doi: 10.1155/2024/8813121. eCollection 2024. PMID 40225925
- [Derived] Cechova A, Honzik T, Edmondson AC, Ficicioglu C, Serrano M, Barone R, De Lonlay P, Schiff M, Witters P, Lam C, Patterson M, Janssen MCH, Correia J, Quelhas D, Sykut-Cegielska J, Plotkin H, Morava E, Sarafoglou K. Should patients with Phosphomannomutase 2-CDG (PMM2-CDG) be screened for adrenal insufficiency? Mol Genet Metab. 2021 Aug;133(4):397-399. doi: 10.1016/j.ymgme.2021.06.003. Epub 2021 Jun 11. PMID 34140212